CLINICAL TRIAL: NCT00398723
Title: Effects of Narrowband UVB Phototherapy on Melanocyte Proliferation in Patients With Vitiligo
Brief Title: Narrowband UVB Treatment in Patients With Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Sullivan-Whalen (Other)
Responsible Party: Sponsor-Investigator, Mary Sullivan-Whalen, Co-Investigator, Rockefeller University
Organization: Rockefeller University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUH IRB # JCO 0590
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Vitiligo
Keywords: Narrowband UBV Phototherapy; Skin biopsies
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitiligo (Experimental): adult patients (age 18 or greater) with extensive vitiligo warranting treatment with whole body NB-UVB
  Interventions: Device: Narrowband UVB

INTERVENTIONS:
Device: Narrowband UVB — Treatment three to seven times weekly for a total of 12 to 26 weeks (36 to 168 treatments). Dosing of NB-UVB will begin at 100-280 mJ/cm2, depending on tolerance and skin type, and will be titrated 10-20% per session until clinical efficacy or symptomatic erythema

SUMMARY:
The study offers narrowband UVB light therapy to patients who have 5% of their body involved with vitiligo.

The hypothesis is that Narrowband UVB promotes melanocyte proliferation in vitiligo lesions.

DETAILED DESCRIPTION:
All patients will receive phototherapy, with narrowband UVB, three times a week for six months, or a total of 78 treatments. 6mm punch skin biopsies (2) will be done prior to starting therapy, once during treatment (2) and at the completion of the study (2). Clinical assessments and photography will be done parallel to the skin biopsies. Results (clinically and histologically) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or greater
* Vitiligo with extensive skin involvement (>5% body surface affected).

Exclusion Criteria:

* No treatment with topical steroids, calcineurin inhibitors or vitamin D analogs for at least 4 weeks prior to entering the study.
* No treatment with systemic therapies, including methotrexate, etretinate, PUVA, or cyclosporine 4 weeks prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number of melanocytes per unit length of skin surface | pre-treatment, early repigmentation, 75% repigmentation of total body

SECONDARY OUTCOMES:
Clinical improvement | first visit and last visit

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States